CLINICAL TRIAL: NCT03974529
Title: Intensive Running Exercise Improves Parkinson's Motor and Non-motor Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Danny Tat Ming Chan, Head of Neurosurgery, Principal Investigator, Honorary Clinical Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Run for PD -v1; NTEC-2018-0330 (Registry Identifier: Joint CUHK-NTEC Clinical Research Ethics Committee (CREC))
Record Dates: First submitted 2019-04-17; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease
Keywords: Intensive running; Gait; Balance; Motor symptoms of Parkinson's disease; Non-motor symptoms of Parkinson's disease; UPDRS score; Physiotherapy; Quality of life
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled single-blinded study. 30 patients will be included and randomized to intervention arm or control arm in a ratio of 2 to 1. Informed consent will be signed after the patient is fully informed about the procedures and prior to the baseline assessments.
  Intervention arm
  * Number of participants: 20
  * Venue: Shatin playground
  * Supervisors: licensed coaches (2 to 4 per session)
  * Training session: 30 minutes of warm-up stretching + 60 minutes supervised progressive aerobic endurance track running
  * Targeted intensity: 60-75% of maximum heart rate (HR max = 220 - age) OR 40-50% heart rate reserve (HRR= HR max - HR rest)
  * Frequency and training period: 2 sessions per week, for 24 weeks
  Control arm
  * Number of participants: 10
  * Venue: Indoor gymnasium
  * Supervisor: a physiotherapist
  * Training session: 60 minutes of physical stretching
  * Frequency and training period: 1 session per week, for 24 weeks
Who Masked: Outcomes Assessor
Masking Description: The assessment will be taken by three blinded assessors (one occupational therapist, a registered research nurse and a research assistant) at baseline, at completion of the training and 6 months after, at Prince of Wales Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive running arm (Experimental): 20 patients will be assigned randomly to intensive running arm (intervention arm). They will be required to complete a designed training protocol.
  Interventions: Behavioral: Intensive running
- Physiotherapy arm (Active Comparator): 10 patients will be assigned randomly to physiotherapy arm. They will be required to complete a designed training protocol.
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Intensive running — The patients who are assigned to this group will be required to finish a 90 minutes of training protocol, containing 30 minutes' warm-up stretching, and 60 minutes of supervised progressive aerobic endurance track running. The training takes place two time per week, for 24 weeks.
  Arms: Intensive running arm
Behavioral: Physiotherapy — The patients who are assigned to this group will be required to finish a 60 minutes of physiotherapy session. The training takes place once per week, for 24 weeks.
  Arms: Physiotherapy arm

SUMMARY:
High quality clinical trial and meta-analysis have demonstrated short term, and to a lesser extent, long term benefits in various outcome measures. To achieve positive effects, supervised progressive strength and aerobic endurance training program of 12 weeks was required. Extended progressive strength training improved muscle strength for up to 24 months. While aerobic endurance training would increase walking capacity up to 16 months. 1 There are data suggesting a threshold of intensity of exercise to be reached for the positive effect. This overall body of evidence suggests that regular vigorous exercise should be accorded a central place in the treatment of Parkinson's disease.

However, there was no evidence about regular intensive exercise of running in Parkinson's disease. And most of the studies were not randomized with a control group.

In this study, the investigators are to investigate the effect of regular vigorous aerobic exercise training of running on motor and non-motor symptoms, and quality-of-life of people with Parkinson's disease.

DETAILED DESCRIPTION:
There is growing volume of evidences support the positive effect of exercise and physical therapy to Parkinson's disease. Various exercise types have shown different positive effects. Gait training for 4 weeks showed a moderate improvement in balancing while balance training of 8 to 26 weeks decreased fall rate. Cued exercise would mildly increase the speed of the gait. Complementary exercises, such as Tai Chi and dancing, have shown improvement in balancing of the patients.

One of the main complaints of Parkinson's disease is rigidity. It is because of the musculoskeletal impairments which compromise the flexibility and stability of both axial structure (spine) and the extremities. Truncal stiffness and rigidity results in a stooped posture, which further undermines one's balance and agility. Flexibility training (stretching) is shown to be beneficial to all stages of patients with Parkinson's disease, in terms of improved both range of movement in joints and spinal stability. It is recommended that regular stretching should be the first step in one's exercise program to combat the muscle rigidity. High quality clinical trial and meta-analysis have demonstrated short term, and to a lesser extent, long term benefits in various outcome measures. To achieve positive effects, supervised progressive strength and aerobic endurance training program of 12 weeks was required. Extended progressive strength training improved muscle strength for up to 24 months. While aerobic endurance training would increase walking capacity up to 16 months.

There are data suggested a threshold of intensity of exercise to be reached for the positive effect. This overall body of evidence suggests that regular vigorous exercise should be accorded a central place in the treatment of Parkinson's disease.

In this study, the investigators are to investigate the effect of regular vigorous aerobic exercise training of running on motor and non-motor symptoms, and quality-of-life of people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with idiopathic Parkinson's disease, aging from 40 years to 60 years old.
2. Patient who are able to walk independently without walking aids for a distance of 30 meters.

Exclusion Criteria:

1. Previous history of other neuro-degenerative diseases
2. Presence of ischemic heart disease or musculoskeletal and cardiopulmonary diseases
3. Presence of physical disability
4. History of regular running practice in the past 6 months.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-29 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's disease rating scale Overall Score | Six months after finishing the training
  A comprehensive 50 question assessment of both motor and non-motor symptoms associated with Parkinson's. The MDS-UPDRS features sections that require independent completion by people affected by Parkinson's and their carers, and sections to be completed by the clinician.
  Part 1: non-motor experiences of daily living Part 2: motor experiences of daily living Part 3: motor examination Part 4: motor complications. Some sections of the UPDRS scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).
Parkinson's Disease Questionnaire - 39 (PDQ39) Quality of Life Score | Six months after finishing the training
  The PDQ39 is a 39-item self-reporting questionnaire which assess the Parkinson's disease associated health related quality over the last month. PDQ-39
  There are 39 questions in the long form Parkinson's Disease Questionnaire, with 8 discrete scales:
  mobility (10 items) activities of daily living (6 items) emotional well-being (6 items) stigma (4 items) social support (3 items) cognitions (4 items) communication (3 items) bodily discomfort (3 items) Patients are asked to think about their health and general well-being and to consider how often in the last month they have experienced certain events (e.g. difficulty walking 100 yards). Patients are asked to indicate the frequency of each event by selecting one of 5 options (likert Scale): never/occasionally/sometimes/often/always or cannot do at all.

SECONDARY OUTCOMES:
Endurance | Six months after finishing the trainingBaseline, one month after finishing the training, and six months after finishing the training
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. It is suitable in assessing endurance in patients with Parkinson's disease
Gait performance | Six months after finishing the training
  Fastest walking speed: Duration for individual walks without assistance for 10 meters
MiniBest Test Score | Six months after finishing the training
  MiniBest test is an evaluation system focusing on the balance of patients with Parkinson's disease. The maximum score for the system is 28 whereas the minimum score is 0. The higher the score is, the better the patient's function.
Mood | Six months after finishing the training
  Symptoms related to anxiety and depression measured with Anxiety and depression Hospital Anxiety and Depression Scale (HADS). It is a commonly used tools in hospital settings to determine the level of depression and anxiety. There are 14 questions in total, with 7 items assessing level of depression whereas 7 for the level of anxiety. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the higher level of depression/ anxiety patient is experiencing.The HADS uses a scale and therefore the data returned from the HADS is ordinal.

CONTACTS AND LOCATIONS:
Overall Officials: Danny TM Chan, Dr., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Patient do not consent for sharing the data.

REFERENCES:
- [Background] Mak MK, Wong-Yu IS, Shen X, Chung CL. Long-term effects of exercise and physical therapy in people with Parkinson disease. Nat Rev Neurol. 2017 Nov;13(11):689-703. doi: 10.1038/nrneurol.2017.128. Epub 2017 Oct 13. PMID 29027544
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: Key Citation PARKINSON ' S DISEASE A Comprehensive Approach to Exercise — https://insights.ovid.com/crossref?an=00135124-201107000-00006
- See also: Key Citation: Parkinson's disease: fitness counts — http://www.parkinson.org/sites/default/files/Fitness_Counts.pdf

DOCUMENTS (2):
  • Study Protocol (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03974529/Prot_000.pdf
  • Informed Consent Form (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03974529/ICF_001.pdf